CLINICAL TRIAL: NCT03555331
Title: Intervention Nurses Start Infants Growing on Healthy Trajectories (INSIGHT) - Long Term Follow-Up
Acronym: INSIGHT
Status: Completed | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Penn State University (Other); National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University at Buffalo (Other); University of Connecticut (Other)
Responsible Party: Principal Investigator, Ian M. Paul, MD, Professor of Pediatrics and Public Health Sciences; Chief, Division of Academic General Pediatrics; Vice Chair of Faculty Affairs, Department of Pediatrics, Milton S. Hershey Medical Center
Other Study IDs: STUDY000034493; R01DK088244 (NIH)
Record Dates: First submitted 2018-06-01; First posted 2018-06-13 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Child Obesity
Keywords: responsive parenting
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- INSIGHT participants: Mother-child dyads who enrolled in the INSIGHT Study and participated from early infancy to age 3 years will be followed through age 9 years.
  Interventions: Behavioral: Child Safety Control Intervention; Behavioral: Responsive Parenting Intervention

INTERVENTIONS:
Behavioral: Child Safety Control Intervention — In the study period which spanned from early infancy through age 3 years, the child safety intervention group was given an educational program with messages focused on child and home safety, guided by the American Academy of Pediatrics and the Academy's guide for health supervision, Bright Futures. The observation-only study extension will not include any intervention, rather it will assess any long term outcomes from the education given to parents when their children were 0-2 years old.
Behavioral: Responsive Parenting Intervention — During infancy, the Responsive Parenting group was given an educational program containing messages providing developmentally appropriate guidance to parents of infants on responsive parenting and healthy lifestyle aimed at preventing rapid weight gain in infancy and overweight at age 3 years. The new study period will not include any intervention, rather it will assess any long term outcomes from the education given to parents when their children were 0-2 years old.

SUMMARY:
Intervention Nurses Start Infants Growing on Healthy Trajectories (INSIGHT 2)-Long Term Follow-up will follow participants enrolled in the Intervention Nurses Start Infants Growing on Healthy Trajectories (INSIGHT) (NCT01167270) study from age 3 years through the developmentally important time at school-entry around age 6 years and into middle childhood at age 9.

DETAILED DESCRIPTION:
INSIGHT(NCT01167270) is a randomized, clinical trial evaluating a responsive parenting (RP) intervention designed to prevent rapid infant weight gain and childhood obesity among first-born infants. RP has been shown to promote a range of adaptive outcomes in children including secure attachment, cognitive development, and self-regulation of emotions and behavior with the potential for many beneficial effects including obesity prevention. INSIGHT's RP intervention is being compared with a home safety control intervention using a birth cohort of 279 infants and parents who received four home visits during the first year followed by annual clinic visits through age 3 years.

The study team will now follow the INSIGHT cohort with growth measurements from ages 5-9 years and with an in-depth assessment of parenting and child behaviors around the time of grade school entry at age 6. The study extension is observational and participants will not be given any further parenting or safety guidance as described in the initial grant.

ELIGIBILITY:
Inclusion Criteria:

* Participating in the INSIGHT study.

Exclusion Criteria:

* Unwilling to continue study participation for the study continuation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: INSIGHT had a birth cohort of 279 infants and parents. Participating dyads received four home visits during the first year followed by annual clinic visits through age 3 years. This study extension will include actively participating parents and children from this original birth cohort that are willing to continue to be followed by the study team.
Sampling Method: Non-Probability Sample
Enrollment: 216 (Actual)
Dates: Start 2018-06-07 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
Efficacy of an early life responsive parenting (RP) intervention as demonstrated by a main effect for study group on BMI from ages 3 through 9 years | 6/2018 through 9/2024
  Repeated measures ANOVA will be used to examine BMI change from ages 3 through 9 years, testing for persistence of the RP effect across time points, and also for an interaction between occasion and intervention group. Tests for an interaction between child sex and study group will be performed.

SECONDARY OUTCOMES:
Mean BMI z-score | 6/2018 through 9/2024
  ANOVA at ages 5, 6, and 9 years.
Proportion in each group overweight (BMI >=85th percentile) or obese (BMI >=95th percentile) | 6/2018 through 9/2024
  Logistic regression analysis will be used to examine the intervention effects on the overweight/obese outcomes at 5, 6, and 9 years.
Test the sustained efficacy and long-term effects of an early life responsive parenting (RP) across the study period | 6/2018 through 9/2024
  Repeated measures ANOVA will be used to examine BMI change from ages 3-4 weeks through 9 years.

CONTACTS AND LOCATIONS:
Overall Officials: Ian M Paul, MD, MSc, Principal Investigator — Penn State Hershey Milton S Hershey Medical Center; Jennifer Savage, PhD, Principal Investigator — Penn State University
Locations (2):
- United States (2):
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Penn State University, State College, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Paul IM, Williams JS, Anzman-Frasca S, Beiler JS, Makova KD, Marini ME, Hess LB, Rzucidlo SE, Verdiglione N, Mindell JA, Birch LL. The Intervention Nurses Start Infants Growing on Healthy Trajectories (INSIGHT) study. BMC Pediatr. 2014 Jul 18;14:184. doi: 10.1186/1471-2431-14-184. PMID 25037579
- [Derived] Paul IM, Barton JM, Anzman-Frasca S, Hohman EE, Buxton OM, Hess LB, Savage JS. Long-Term Effects of a Responsive Parenting Intervention on Child Weight Outcomes Through Age 9 Years: The INSIGHT Randomized Clinical Trial. JAMA Pediatr. 2025 Aug 1;179(8):827-835. doi: 10.1001/jamapediatrics.2024.6897. PMID 40063048